CLINICAL TRIAL: NCT04091711
Title: Clinical Study to Evaluate the Safety, Usability and Efficacy of the ReX-C® System in Measurement and Management of Medication Adherence and Clinical Self-reporting, in Oncology Patients Receiving Home-based Oral Oncolytic Therapy
Brief Title: Evaluation of ReX-C® System for Medication Adherence in Oncology Patients Taking Oral Oncolytics
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting next model of the device
Sponsor: Dosentrx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXC-034-2019-CLE
Record Dates: First submitted 2019-09-09; First posted 2019-09-17 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Oncology; Adherence, Medication; Side Effect
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Open study for subjects receiving home-based oral oncolytic treatment. Subjects receive these medication by ReX-C device. Medication adherence, treatment instructions and side effects are recorded and monitored online in real time during the Study, by the ReX-C system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ReX-C intervention (Experimental): Subjects use ReX-C to receive oral oncolytic medications. Adherence data, side effects and response to treatment are monitored online in real time via ReX-C cloud.
  Interventions: Device: ReX-C system

INTERVENTIONS:
Device: ReX-C system — Oral oncolytic medications are dispensed to patients via ReX-C system

SUMMARY:
In recent decades, an increasing number of oral anticancer medications (oral oncolytics) have been approved. Oral oncolytics now make up to 30% of the oncology market, and their use is continually expanding.

Oral oncolytics can be a significant benefit for patients and providers. Patients who receive them often report a greater sense of control over their treatment, less interference with daily work and social activities, reduced travel time and costs, and the elimination of discomfort associated with an IV line. In rural areas, the oral route is crucial because the closest treatment center may be hours away and weather may complicate travel. Moreover, oral therapy is less invasive and reduces nursing time in infusion suites and risks to patients.

However, making cancer treatments available in oral form transfers most of the responsibility for correct administration of the drug to the patient. The more complex the oral treatment regimen, the higher the risk of errors and non-adherence. Oral Oncolytics are high-risk and high cost drugs. Hence, with this transfer of responsibility comes the need to support patients in their adherence to the directed regimen and to effectively monitor them at home.

DETAILED DESCRIPTION:
ReX is a hand-held, mobile device intended to provide solid oral medication on patient demand according to a pre-programmed treatment protocol. ReX addresses poor patient adherence, tracks patient's response to treatment and enhances patient engagement to therapy. The system comprises a reusable drug dispensing unit (Dispenser), a disposable Cassette containing the prescribed medication, a cellphone app, and the ReX cloud. The Dispenser manages pill administration. It includes a touch screen which guides the user and presents patient-specific clinical surveys and therapy information. The Dispenser contains a chargeable battery and indicators demonstrating device and battery status; a pill window enabling pills to be viewed; operational sensors; and communication to an app on cellphones. The patient receives the Cassette from the pharmacy, pre-filled with his/her specific medication. The Cassette is inserted into the Dispenser where it is locked in place. All therapy and patient survey data are transferred to a patient-specific domain on DosentRx' proprietary web-based cloud, named Dose-E®.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, at least 18 years of age
2. Subject is able to swallow pills and during training successfully achieves 2 administrations of "demo" pills (Tic-Tac mints) by the ReX-C.
3. Subject is able to read and understand the Informed Consent Form.
4. Subject was diagnosed with cancer and receives oral oncology medication.
5. Subject is intended to receive Afinitor OR Sutent OR Lenvima during the 2 months study period.
6. Subject takes medication therapy at home.
7. Subject is fluent in one of the following languages: Hebrew, English, Russian, Arabic.

Exclusion Criteria:

1. Subject has physical or mental disabilities which prevents their enrolment in this study, such as poor fine motor skills, impaired visual or auditory faculties, mental disorders or other impairment affecting ability to provide Informed Consent or use the ReX-C dispensing unit effectively.
2. Subject failed to extract 2 Tic-Tacs with the Rex-C device during training.
3. Subject is participating in another clinical study that does not permit participation in two studies simultaneously.
4. Subject is at end stage or terminal illness with anticipated life expectancy of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Number of safety events during administration of oral oncolytic medications by ReX-C | 8 weeks
  Safety events include: pill overdose, pill inhalation during pill ingestion, pill malformation upon dispensing and any severe adverse events related to pill intake by the ReX-C device.
Rate of subjects feel comfortable to use ReX-C for pill intake and side effects report | 8 weeks
  At least 70% of subjects: -
  * Complete the duration of the study with Rex-C.
  * Define the system as comfortable to use and are willing to continue using it for their oncolytic medication treatment.
Rate of adherence (number of pill intakes) during treatment with ReX-C | 8 weeks
  * Up to 90% of pills are taken as prescribed
  * At least 80% of subjects follow treatment instructions, and response to ReX-C reminders and alerts.
Rate of monitoring subjects' home-based treatment by the clinical staff and satisfaction of the clinical team | 8 weeks
  At least 80% of clinical team:
  * are satisfied with the use of the system and report that it is beneficial in monitoring patients' adherence and response to treatment.
  * report that the system facilitates better communication with the patient and provides more appropriate real-time response compared to routine care.
  * are interested in integrating the system into the oncology department for routine administration of home-based medication for oncology patients.

SECONDARY OUTCOMES:
Number of actual pill intakes by ReX-C system, compared with the number of prescribed pills | 8 weeks
  Test if the number of pills prescribed and given to the subjects is higher than that actually taken during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Geva, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Oncology Unit, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No